CLINICAL TRIAL: NCT03625349
Title: Passive Limb Movement: A Tool to Assess Vascular Health and Guide Rehabilitation
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: E3207-R; E1697-R (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2018-07-24; First posted 2018-08-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Aging; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — omega-N-Methylarginine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PLM participants: Participants who undergo passive leg movement, with and without LNMMA.
  Interventions: Drug: NG-Monomethyl-L-Arginine

INTERVENTIONS:
Drug: NG-Monomethyl-L-Arginine — Inhibitor of nitric oxide synthase.
  Other Names: LNMMA

SUMMARY:
Brief Summary:

Current U.S. Veteran demographics reveal an aging population with significant cardiovascular dysfunction. This ultimately manifests as mobility limitation, inactivity, and a subsequent worsening of cardiovascular disease (CVD) that often leads to death. However, despite this clear negative cycle of events, there is not a single clinically accepted, and therefore routinely utilized, method of assessing vascular health. As nitric oxide (NO) is anti-atherogenic and cardioprotective, identifying an in vivo bioassay of NO bioavailability has significant worth in this arena. Fueled predominantly by the VA Merit Award prior to this renewal application, single passive leg movement (sPLM) and the subsequent blood flow increase, measured non-invasively by ultrasound Doppler in the common femoral artery, is emerging as a method by which vascular endothelial function and therefore NO bioavailability can be determined. However, although this work has yielded an initial characterization of sPLM and established this method to be a novel, valid, and a clinically relevant approach to determine vascular health, further understanding of the sPLM response with advancing age and, ultimately, its implementation and assessment in both rehabilitation and clinical arenas is still necessary. With the growing interest in personalized medicine, the development of tools, such as sPLM, that allow individualized assessments to guide the physician, the patient, and the rehabilitative team, are essential. Therefore, two specific aims are proposed that will address the Central Hypothesis that the sPLM paradigm provides a clinically meaningful assessment of endothelial function. First, cardiac rehabilitation will be assessed by sPLM in the elderly, and, coupled with studies in the young, will elucidate the predominant pathways responsible for the change in endothelial function with aging and rehabilitation. Second, the CVD diagnostic value of the sPLM assessment of endothelial function will be evaluated relative to classic measures and markers of subclinical disease in order accelerate the inclusion of endothelial dysfunction as a CVD risk factor. The proposed studies aim to catalyze the transition of the assessment of endothelial function by sPLM from research to clinical practice.

DETAILED DESCRIPTION:
Importance and impact: It is becoming increasingly apparent that arterial endothelial dysfunction contributes significantly to the age-related downward spiral that includes mobility limitation, frailty, and ultimately cardiovascular disease (CVD). Endothelial dysfunction has been documented to manifest in the coronary epicardial and resistance vasculature as well as the peripheral arteries, indicating that such dysfunction is a systemic condition. Indeed, there is a growing appreciation that the vast majority of CVD is, in fact, associated with endothelial dysfunction. Thus, developing a better understanding of the relationship between arterial aging and CVD is one of the most important clinical challenges that we currently face. The vascular endothelium, a single layer of cells lining the blood vessel wall, plays an essential role in maintaining both arterial function and health. In either an autocrine or paracrine fashion, vascular endothelial cells synthesize and release numerous biologically active molecules that modulate arterial structure as well as vasodilatory, thrombolytic, and vasoprotective functions. The important role that nitric oxide (NO) plays in vasodilation. The transition from normal endothelial function to the phenotype of endothelial dysfunction contributes to the development of atherosclerosis and increased CVD risk. Specifically, these vascular changes, catalyzed by diminished NO bioavailability, lead to vasoconstriction and an endothelial state that is pro-coagulative, pro-proliferative, and pro-inflammatory. The recognition that the endothelium is not simply a passive interface between blood and vessel wall, but is also the site of NO production, has led to great advances in the field of vascular research. Indeed, endothelial-derived NO is now not only recognized as one of the most important vasodilators, particularly in the muscular arteries, but it also is apparent that NO inhibits other key events associated with the development of atherosclerosis, such as leukocyte adhesion and migration, platelet adhesion and aggregation, and smooth muscle cell proliferation. Thus, attenuated NO bioavailability is evidence of a broadly dysfunctional endothelial phenotype, and, therefore, the assessment of NO-mediated vasodilatory capacity provides significant insight into the integrity and function of the endothelium. Although the process of CVD can begin early in life and is accelerated by the aging process, endothelial dysfunction, a recognized precursor to atherosclerosis, precedes the structural changes associated with this disease and so can be used as a predictor of CVD onset.

Originality: Most, if not all, CVD risk factors are associated with endothelial dysfunction, and risk factor modification can lead to improved endothelial function. With the growing interest in personalized medicine, the development of diagnostic tools, that allow individualized assessments of endothelial function to guide the physician, the patient, and the rehabilitative team, are essential. However, although, over the past 20 years, several methodologies have been developed to assess endothelial function in humans, and these approaches have contributed extensively to clinical research, none have been adopted into clinical practice. In fact, not a single method for assessing endothelial function has been recommended by clinical guidelines for the diagnosis of CVD and the guidance of prevention strategies for primary or secondary CVD. From work performed in the current Merit Review Award, the novel single passive leg movement (sPLM)-induced increase in leg blood flow (LBF) approach to assess endothelial function appears to be the clinically relevant tool that has long been missing from the healthcare provider's arsenal. However, the additional studies proposed in this renewal application are needed to confirm this conclusion, especially as it relates to rehabilitation. Importantly, the sPLM paradigm can guide rehabilitation in several ways. First, the high diagnostic value would provide earlier detection of CVD risk, particularly as endothelial dysfunction precedes many of the other risk factors, and the sPLM testing can be used to recommend and motivate patients to undergo rehabilitation. Second, the sPLM assessment can be used to determine the efficacy of rehabilitation in order to guide program development. If rehabilitation is not improving vascular function, the program can be modified to address this CVD risk factor, with the impact on other outcomes in mind. Third, the sPLM paradigm can be used more acutely throughout a rehabilitation program to provide "real-time" feedback about endothelial function, allowing practitioners to personalize the program for each patient, again with other outcomes in mind.

Contribution to Veterans Health Administration (VHA): VA demographics reveal a population that is significantly skewed toward the older sector and, thus, heavily burdened by age-associated CVD. Even in the population at large, it is estimated that by the year 2050 over 21% of people will be over 60 years of age. Although these data are impressive, the Veteran population is far ahead of these predictions with 51% (12.3 million) of Veterans already over 60 years of age. As advancing age is the major risk factor for CVD, the risk of CVD increases progressively across the lifespan and although death rates as a result of CVD have fallen over the last 50 years, CVD remains the leading cause of morbidity and mortality in the U.S. Given the already accelerated aged demographics in the VA Health Care System and the strong link between CVD and age, there is little doubt that the burden of CVD-related healthcare costs within the VA will continue to grow. Thus, it is not surprising that aging and mobility limitation, both of which are linked to endothelial dysfunction, are two priority areas emphasized by the VA RR&D Service and are Medical Research Priorities for the VHA system as a whole.

Post cuff-occlusion flow-mediated vasodilation (FMD) as a test of NO bioavailability: Prior to our development of the novel sPLM approach to assess endothelial function, fueled predominantly by the current Merit Review Award, perhaps the most likely method to be adopted for routine clinical use was the post cuff-occlusion FMD test, typically performed in the brachial artery. In 1992, Celermajer et al. introduced this method of measuring the changes in conduit artery diameter following a period of circulatory occlusion as a non-invasive approach for in vivo determination of endothelium-dependent vasodilation in humans. In the more than two decades that have followed, the application of FMD testing in clinically-based research has become widespread, a progression that is exemplified by the adoption of this methodology into large-scale clinical trials, including recent phases of the Framingham Heart Study. The FMD test is particularly appealing due, at least in part, to a previous report revealing a weak correlation between vasodilatory capacity of the peripheral and coronary arteries, implicating FMD as a potential surrogate measure of coronary endothelial health. Further, it has been clearly demonstrated that FMD provides independent predictive information for future cardiovascular events beyond traditional risk factors. FMD testing has, thus, emerged as a non-invasive approach for determining vascular function in health and disease. However, predominantly due to several methodological deficiencies and significant challenges in terms of implementation, FMD has never been embraced as a clinical tool. Perhaps one of the most attractive aspects of FMD testing is that it has been purported to provide an assay of vascular endothelial NO bioavailability. As the presence of this endothelially-derived vasodilator has become synonymous with vascular health, the prospect of quantifying NO in a non-invasive manner makes FMD testing particularly appealing for both risk assessment and patient prognosis. The ability of NO synthase (NOS) inhibition with LNMMA (NG-monomethyl-L-arginine) to completely abolish radial and brachial artery FMD provided initial evidence that FMD is governed primarily through the release of NO. However, in the face of significant technical and methodological refinements in the field, recent studies challenge the existing dogma regarding the NO dependent nature of the FMD response. Indeed, the two most recent studies in the radial artery have identified only a minimal (0-33%) reduction in FMD after the administration of LNMMA, a NOS blocker, leaving considerable uncertainty as to whether this test can still be relied upon to provide an assay of NO bioavailability. Indeed, our group, using up-to-date measurement techniques and the typical site of assessment (brachial artery), demonstrated that the majority of vasodilation provoked by brachial artery FMD testing is not attributable to NO. In fact, the intra-arterial delivery of L-NMMA resulted in only a modest ( 33%) reduction in FMD. Critically, L-NMMA administration also reduced the post-occlusion hyperemic response, thereby diminishing the shear stimulus for brachial artery vasodilation. When this effect was taken into account, FMD normalized for shear rate was not different between control and L-NMMA conditions. Additionally, changes in FMD are highly dependent upon assessing very small changes in artery diameter. Furthermore, FMD transiently increases with exercise training over the initial 4 weeks, but returns to pre-training values by the 8th week due to arterial remodeling. This plasticity in diameter greatly limits the use of FMD as a diagnostic assessment in clinical and rehabilitation arenas. Finally, although FMD has been demonstrated to correlate with CVD risk, it provides only marginal diagnostic value for CVD. These findings add to the growing uncertainty surrounding the interpretation of FMD test results, the usefulness of this approach clinically, and emphasize the need to develop a new and clinically relevant tool to assess endothelial function and NO bioavailability.

sPLM as a test of NO bioavailability: Originally, our group and others focused on the peripheral and central hemodynamic responses to sPLM, and its previous variants, as a reductionist model to better understand the factors controlling movement-induced hyperemia. By removing the increase in metabolism associated with active exercise, important findings related to the control of skeletal muscle blood flow were revealed. Specifically, in healthy humans, following the initial onset of passive movement, there is a transient, yet robust, increase in LBF. Through various experimental approaches we have characterized the roles of afferent feedback, the muscle pump, perfusion pressure, cardiac innervation/denervation, and age in the sPLM response. However, most germane to this Merit Review renewal application, funded by the current Merit Review Award, we have determined the role NO plays in the sPLM-induced blood flow response in both young and old subjects. At rest, NOS inhibition has consistently been documented to decrease limb blood flow and vascular conductance by 30 to 40%, indicating an essential role of NO in controlling basal blood flow. During active exercise, the reduction in blood flow following NOS inhibition is typically less than at rest, falling in the range of 5 to 25%.This implies a reduced contribution of NO to exercise-induced hyperemia, an experimental paradigm characterized by increased metabolism, which also likely plays a significant role in elevating blood flow during exercise. In contrast, the sPLM-induced hyperemia, which does not evoke a peripheral metabolic response, is intuitively more likely to be predominantly NO-mediated. Indeed, in young healthy subjects the inhibition of NOS, with an intra-arterial L-NMMA infusion in the passively moved leg, revealed that NO contributes to 65-80% of the hyperemia and vasodilation associated with sPLM. In contrast, there was minimal effect of L-NMMA in the old. The sPLM response is also markedly attenuated in old, compared to young, subjects. Substantial evidence supports NO bioavailability is low in old subjects and, as sPLM is highly NO-mediated, both the diminished sPLM response and diminished effect of L-NMMA are consistent with such diminished NO bioavailability. This supports the sPLM as a good assessment of endothelial function because it tracks physiological differences across populations. This robust and easily measured reduction in NO-mediated vasodilation and subsequent hyperemia suggests that sPLM induced blood flow has significant promise as a new approach to assess NO-mediated endothelial function, an important predictor of CVD risk, and could be an important tool to assess rehabilitation.

sPLM and FMD directly compared: Being noninvasive and with evidence of mirroring coronary endothelial function to some degree, FMD is by far the most common approach to assess vascular function in clinical research and has been in existence for over 20 years. However, FMD testing can be a somewhat capricious endeavor exhibiting significant operator dependency, difficulty with performance, a reliance upon very small vessel diameter changes (typically less than 0.4 mm), uncertainty about how to account for varying shear stimuli, and concerns regarding reproducibility, all of which combine to explain why FMD has yet to be adopted clinically. Moreover, and of real significance, the diagnostic value of FMD for CVD is only marginal and inconsistent. In a relatively recent article, highly germane to this proposal, published in the Contemporary Reviews in Cardiovascular Medicine section of the journal Circulation, Flammer et al. discuss many of these issues in their article entitled "The assessment of endothelial function: from research to clinical practice". Interestingly, they conclude that a clinical tool to assess endothelial function, suitable for daily practice has yet to be established. Of note, sPLM was not mentioned in this review for, at this time, this novel method was truly in its infancy.

sPLM, aging and NO: It is well recognized that endothelial function and, therefore NO bioavailability is attenuated with age and, therefore, if sPLM is, indeed, a good indicator of endothelial function, it would be anticipated that the role of NO would be diminished in the elderly population. Funded by the current VA Merit Review Award, we have confirmed this supposition utilizing the sPLM assessment of endothelial function. Specifically, we have documented that in young healthy subjects, the inhibition of NOS by L-NMMA reduced the hyperemic response to sPLM, as assessed by leg blood flow area under the curve (AUC), by 65-80%. In contrast, in old subjects (>70 yr.), compared to their young counterparts, there was a greatly attenuated sPLM-induced hyperemia in the control condition (AUC 24 vs 147 ml) and a nonsignificant effect of NOS blockade, both of which are consistent with a diminished NO bioavailability. These findings confirm that endothelial function is diminished with age and this can be explained by a reduction in NO bioavailability, both of which can be documented by the use of sPLM.

sPLM as a valid screening test for age-related endothelial dysfunction: During the current VA Merit Review Award, in healthy young and old subjects, we documented that the peripheral hemodynamic response to sPLM provides a highly sensitive and specific assessment of the recognized age-related fall in endothelial function. Compared to young subjects, the LBF response to sPLM in the old was markedly attenuated. sPLM LBF AUC revealed a clear delineation between young and old, with a cut-score of 60 ml. These data document the capacity for the peripheral hemodynamic responses to sPLM to provide clear and potentially diagnostic information to facilitate the classification of an individual as exhibiting, or not, age-related endothelial dysfunction, which is currently missing as a CVD risk factor. Additionally, these findings revealed that, in young and old populations, the relatively easy to assess, LBF AUC, alone, is an appropriate surrogate for the more complex leg vascular conductance which requires the simultaneous assessment of beat by beat blood pressure. Therefore, the hyperemic response to sPLM exhibits the prerequisite qualities of a valid screening test for peripheral endothelial dysfunction, as evidenced by an sPLM assessed endothelial function, CVD risk, and physical activity: There is significant evidence that endothelial dysfunction is associated with CVD risk. In fact, the more risk factors that are present, the worse are both the epicardial56 and peripheral endothelial function. Endothelial dysfunction may, therefore, represent the effect of these risk factors on vascular health. However, it is again important to recognize that impaired endothelial function precedes structural changes and may therefore be considered "a barometer" of the total cardiovascular risk burden of an individual. Thus, even a new method with limited long-term data, which professes to allow the assessment of endothelial function, must demonstrate some relation to CVD risk and risk factor modifications, such as increased physical activity, that can alter CVD risk. Although cross-sectional, there is evidence that endothelial function assessed by the blood flow response to sPLM, is, indeed, attenuated with increasing CVD risk and altered by physical activity. Specifically, although there is variability within each group of subjects, which would be expected and makes individual assessment so important, it is clear that the young and old active subjects exhibit superior endothelial function compared to their age-matched sedentary counterparts, as assessed by sPLM. Additionally, these data suggest that while greater physical activity can improve endothelial function in the old, the elderly subjects do not achieve the same endothelial function of the young subjects, indicating age-related dysfunction. Finally, of apparently healthy subjects, the old inactive subjects have the most attenuated endothelial function due to being male, inactive, and >70 yrs. of age. Of note, in terms of endothelial function, as assessed by sPLM, this group is closest to the patients with heart failure, illustrating the ultimate consequence of numerous CVD risk factors and greatly attenuated endothelial function. This clear link between the sPLM-induced increase in blood flow and CVD risk supports the concept that the development and ultimately the adoption of sPLM as a tool to non-invasively assess endothelial function could have a significant impact on both the VA Health Care System and health care in general. However, currently there are no longitudinal pre- and post-rehabilitation sPLM data to document the efficacy of sPLM in this arena.

In summary, from work performed in the current Merit Review Award, the novel sPLM-induced increase in LBF method to assess endothelial function appears to be both valid, reliable, and clinically relevant. Furthermore, sPLM surpasses previous approaches in many respects, including ease of performance and analysis, is predominantly NO-mediated, and can identify the typical age-related decline in endothelial function with advancing age, apparent inactivity, and disease. sPLM may be the clinically relevant tool that has long been missing from the healthcare provider's arsenal. However, it is now necessary to longitudinally assess sPLM in the rehabilitation arena and to formally assess the diagnostic value, of the sPLM paradigm, for CVD.

Two Specific Aims are proposed, with preliminary data supporting the approach and feasibility.

1. HOW DOES THE PASSIVE SINGLE LEG MOVEMENT (sPLM) ASSESSMENT OF ENDOTHELIAL FUNCTION RESPOND TO CARDIAC REHABILITATION WITH ADVANCING AGE?

   Specific Aim 1A: Determine the impact of cardiac rehabilitation on sPLM assessed endothelial function in both old subjects and patients diagnosed with CVD.

   Approach: sPLM assessments of endothelial function performed in both a group of relatively healthy old subjects and patients diagnosed with CVD before and after a 12 week cardiac rehabilitation program will document the effect of cardiac rehabilitation on endothelial function.

   Hypothesis: The sPLM assessment of endothelial function will improve following cardiac rehabilitation in both relatively healthy old subjects and patients diagnosed with CVD.

   Specific Aim 1B: Determine the predominant vasodilatory pathway responsible for the change in sPLM assessed endothelial function as a consequence of cardiac rehabilitation in old subjects.

   Approach: The measurement of femoral artery blood flow in response to sPLM in young (no rehabilitation) and old subjects (pre- and post-rehabilitation), with and without intra-arterially infused NO synthase (NOS) blockade (NG-monomethyl-L-arginine (L-NMMA)) and in combination with prostaglandin (PG) blockade (Ketorolac) and endothelium-derived hyperpolarizing factor (EDHF) blockade (Fluconazole) will document the role of these dilators in the sPLM response with aging and, subsequently, with cardiac rehabilitation in the old.

   Hypothesis 1: Pre-rehabilitation the old subject's sPLM response will be less dependent on NO and more dependent on PG- and EDHF-induced vasodilation than the young.

   Hypotheses 2: Rehabilitation in the old will increase the role of NO in the sPLM-induced hyperemia, as evidenced by the restoration of the impact of L-NMMA and diminution of the combined effect of PG and EDHF on the sPLM response to that of the young.
2. DOES THE sPLM ASSESSMENT OF ENDOTHELIAL FUNCTION PROVIDE A NOVEL, CLINICALY MEANINGFUL RISK MARKER FOR CVD?

Specific Aim: Determine the diagnostic value of sPLM assessed endothelial function for CVD.

Approach: The sPLM assessment of endothelial function and classic measures (blood pressure, body mass index, fasting blood lipids, and glucose) and markers of subclinical vascular disease (Framingham Risk Score, coronary artery calcium score, ankle brachial index, flow-mediated dilation, carotid intima-thickness, and C-reactive protein) in healthy subjects and patients with CVD will determine the diagnostic value of sPLM for CVD, demonstrating the clinical utility of this measurement.

Hypothesis: The sPLM assessment of endothelial function will have a high diagnostic accuracy for CVD prevalence that is superior to classic measures and markers of subclinical vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy subjects: No evidence of cardiovascular disease.
* Patients undergoing angiography: Clinical referral for an angiography.

Exclusion Criteria:

* Young healthy subjects: Evidence of cardiovascular disease.
* Patients undergoing angiography: Poor kidney function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will range from young healthy volunteers to patients undergoing angiography.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2027-10-29 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Blood Flow Response to passive leg movement. | This outcome measure will be assessed at each study visit through study completion, about 3.5 years.
  Doppler ultrasound will be used to assess movement induced hyperemia in the femoral artery.

CONTACTS AND LOCATIONS:
Overall Officials: Russell S. Richardson, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No